CLINICAL TRIAL: NCT02136121
Title: Prospective Investigation of Robotic Single-port System
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2014-05-05; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Prostate and Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- da Vinci Sp Surgical System (Experimental): da Vinci Sp Surgical System - Robotic - assisted single-port surgery
  Interventions: Device: da Vinci Sp Surgical System - Robotic

INTERVENTIONS:
Device: da Vinci Sp Surgical System - Robotic — robotic assisted laparoscopic single-port system

SUMMARY:
To determine the feasibility of representative urologic procedures as measured by the rate of conversions

ELIGIBILITY:
Inclusion Criteria:

* Prostatectomy:
* Patients age 18-75 years
* BMI <=35 kg/m2
* Confirmed localized adenocarcinoma of the prostate
* Suitable for minimally invasive prostate cancer surgery

Nephrectomy:

* Patient age 18-75 years
* BMI <=35 kg/m2
* Kidney disease amenable to nephrectomy or partial nephrectomy
* Suitable for minimally invasive kidney surgery

Exclusion Criteria:

Untreated active infection (includes local kidney infection)

* Vulnerable population (ex: prisoners, mentally disabled)
* Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions (i.e., cancer)
* Anatomy unsuitable for endoscopic visualization or minimally invasive surgery
* Patient with second primary cancer
* Extensive previous abdominal surgery
* Prior radiation treatment for prostate or kidney cancer
* Patient with distant metastasis
* Complex renal vascular anatomy
* Patient with kidney cancer - stage T3 or N+ M+ **
* Horseshoe kidney**
* Previous ipsilateral kidney surgery **- specific to kidney surgery -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility as measured by the rate of conversions | Intra Operative
  Rate of Conversion to Open approach

SECONDARY OUTCOMES:
Perioperative surgical outcomes | From admission to discharge from the hospital for the primary procedure typically up to 7 days
  Perioperative surgical outcomes length of hospital stay- From admission to discharge from the hospital for the primary procedure
Perioperative Surgical outcomes | Intra-operative
  Rate of Transfusion
Perioperative Surgical Outcomes | 30 day, 1 year , 2 year and 3 year follow up
  Procedure specific wound complications , infection
Post-operative - Continence | 1 year, 2 year and 3 year follow up
  Continence measured by use of pads
Perioperative Surgical Outcome- potency | 1 , 2 and 3 year follow up
  Potency rate administered by International Index of Erectile Function patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Villers, MD, Principal Investigator — Hôpital HURIEZ, CHRU; Jihad Kaouk, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Hôpital HURIEZ, CHRU, Lille, France, France

REFERENCES:
- [Derived] Kaouk JH, Haber GP, Autorino R, Crouzet S, Ouzzane A, Flamand V, Villers A. A novel robotic system for single-port urologic surgery: first clinical investigation. Eur Urol. 2014 Dec;66(6):1033-43. doi: 10.1016/j.eururo.2014.06.039. Epub 2014 Jul 17. PMID 25041850